CLINICAL TRIAL: NCT06397053
Title: Comparison of Robotic Versus Laparoscopic Surgery for Visceral Obesity in Mid-Low
Brief Title: Comparison of Robotic Versus Laparoscopic Surgery for Visceral Obesity in Mid-Low Rectal Cancer: A Propensity-Matched Analysis
Status: Completed | Type: Observational
Sponsor: Daorong Wang (Other)
Responsible Party: Sponsor-Investigator, Daorong Wang, Dr, Northern Jiangsu People's Hospital
Organization: Northern Jiangsu People's Hospital (Other)
Other Study IDs: Visceral Obesity001
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Visceral Obesity; Rectal Cancer; Robotic Surgery
MeSH Terms: conditions — Obesity, Abdominal; Rectal Neoplasms | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laparoscopic surgery with visceral obesity
  Interventions: Procedure: robotic surgery
- robotic surgery with visceral obesity
  Interventions: Procedure: robotic surgery

INTERVENTIONS:
Procedure: robotic surgery — robotic surgery

SUMMARY:
Our team has previously published articles providing detailed descriptions of the steps involved in both RS and LS. All surgeries adhered to the total mesorectal excision (TME) principle. In RS, a surgeon employed the Da Vinci Xi surgical system featuring a five-port setup, while five physicians conducted LS with a similarly configured five-port approach. Both the RS and LS doctors are experienced. The surgeries were conducted according to standard procedures, and the RS group utilized totally robotic rectal resection.

ELIGIBILITY:
Inclusion Criteria:

(1) confirmed pathology of mid-to-low rectal cancer (within 10 centimeters from the anal margin); (2) availability of comprehensive pathological and computed tomography (CT) data; (3) presence of a diagnosis indicating visceral obesity.

Exclusion Criteria:

Multiple tumor

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective investigation included participants who experienced anterior rectal resection using robotic or laparoscopic techniques at the General Surgery Department of Northern Jiangsu People's Hospital between December 2019 and October 2023.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
early postoperative problems | 2019-2023
  early postoperative problems

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No